CLINICAL TRIAL: NCT01107873
Title: Changes of Dorsalis Pedis Artery Flow Pattern After Caudal Block in Children: Observational Study Using a Duplex Sonography
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Hae Keum Kil/Professor, Yonsei University, College of Medicine
Other Study IDs: 4-2010-0085
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-10

CONDITIONS: Anesthesia, Caudal
Keywords: Twenty (ASA status I) unpremedicated children, ages 1 to 5 yr old

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- duplex ultrasonography: conduct duplex ultrasonography after caudal block with sevoflurane anaesthesia in children

SUMMARY:
The purpose of this study is to determine the changes of Dorsalis Pedis Artery Flow Pattern after Caudal Block in Children: Observational Study Using a Duplex Sonography.

ELIGIBILITY:
Inclusion Criteria:

* Twenty (ASA status I) unpremedicated children, ages 1 to 5 yr old, who were scheduled for a day-case urologic surgery

Exclusion Criteria:

* if there were contraindications for caudal block including hypersensitivity to any local anaesthetics, bleeding diathesis, infections at the puncture sites, or pre-existing neurological disease.

Ages: 1 Year to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: children patients who visit Severance hospital
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Investigation of arterial hemodynamics
  Investigation of arterial hemodynamics included peak systolic velocity [PS], end diastolic velocity [ED], mean velocity [MV], time-averaged maximum velocity [TAmax], time-averaged mean velocity [TAmean], pulsatility index [PI], volume flow [VF], and dorsalis pedis artery diameter [D].

CONTACTS AND LOCATIONS:
Overall Officials: Hae Keum Kil, Principal Investigator — Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Korea